CLINICAL TRIAL: NCT05504954
Title: Multilevel Comprehensive HIV Prevention Package for South African Adolescent Girls and Young Women
Brief Title: A Comprehensive HIV Prevention Package for South African Adolescent Girls and Young Women: IMARA SA
Acronym: IMARA-SA pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Desmond Tutu HIV Centre (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Natasha Crooks, Assistant Professor, Human Development Nursing Science, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UG3HD096875 (NIH)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Sexually Transmitted Infection; Hiv
Keywords: HIV prevention; Adolescent girls and young women; South Africa; Mother-daughter intervention
MeSH Terms: conditions — Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Adolescent girl and young women-female caregiver (AGYW-FC) dyads will be randomized to the IMARA-SA intervention arm or a health promotion control arm matched in time and intensity. IMARA-SA and the health promotion program will be delivered as group interventions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMARA-SA intervention arm (Experimental): Participants randomized to the IMARA-SA arm will receive the IMARA-SA intervention (i.e., the intervention group).
  Interventions: Behavioral: IMARA-SA (intervention group)
- Health promotion control arm (Experimental): Participants randomized to the health promotion control arm will receive the health promotion intervention (i.e., the control group).
  Interventions: Behavioral: Health promotion control group

INTERVENTIONS:
Behavioral: IMARA-SA (intervention group) — The IMARA-SA intervention aligns with an ecological framework, emphasizing the intersection of individual, social, and structural determinants of women's sexual health and behavior. Separate FC and AGYW groups run simultaneously and cover parallel content, while joint activities enhance FC credibility as a resource for HIV/STI prevention and facilitate practice of communication skills. Interventionists use interactive and experiential activities. IMARA-SA's goals and motto emphasize strong FC-AGYW relationships, sisterhood, community empowerment, and motivation for HIV prevention, and build group cohesion. FC and AGYW sign a pact to confirm commitment to the program. At the end of Workshop Day 1, participants receive homework to complete during the week. Woven throughout IMARA-SA is the impact of mental health issues, alcohol and drug use, and violence on HIV-risk.
  Arms: IMARA-SA intervention arm
Behavioral: Health promotion control group — The health promotion control intervention is a family-based intervention previously delivered to families in SA and translated into isiXhosa. The intervention promotes healthy living by encouraging good nutrition, exercise, and violence reduction. It will be delivered in the same format as IMARA and will be identical in length and intensity.
  Arms: Health promotion control arm

SUMMARY:
Programs which go beyond individual-level behavior change to reduce HIV and STI infections among adolescent girls and young women in sub-Saharan Africa are essential to meet global HIV targets. Informed, Motivated, Aware and Responsible Adolescents and Adults- South Africa (IMARA-SA) is an evidence-based HIV-prevention intervention for adolescent girls and young women (AGYW) and their female caregivers, which has been adapted for a South African audience. This pilot study will assess feasibility in preparation for a randomized controlled trial (RCT). Additionally, the pilot will examine the preliminary effectiveness of IMARA-SA in reducing sexually transmitted infections (STI) and increasing uptake of HIV testing and counseling (HTC) and pre-exposure prophylaxis (PrEP) at follow-up among AGYW. About 60 AGYW-FC dyads will be enrolled and randomized to IMARA-SA or a health-promotion control arm. Following randomization, the dyads will participate in an ~2-day group workshop (~10 hours), which includes joint and separate mother and daughter activities. AGYW and FC will complete baseline assessments and follow-up assessments approximately 6 months later. Assessments will include surveys, STIs testing (for chlamydia and gonorrhea), and uptake of HTC and a 1-month PrEP prescription. Additionally, the intervention's implementation (e.g., acceptability) will be explored.

ELIGIBILITY:
Inclusion criteria for AGYW include:

1. Black or mixed race;
2. 15-19 years-old;
3. residing in Klipfontein/Mitchells Plain (K/MP);
4. speak isiXhosa or English or a combination of these languages.

Inclusion criteria for FC include:

1. identified by AGYW as a FC;
2. 24 years and older;
3. living with or in daily contact with the AGYW;
4. speak isiXhosa or English or a combination of these languages.

Exclusion Criteria:

AGYW will be excluded from the study if they do not have a FC to participate in the study.

AGYW and FC will be excluded from the study if they:

1. are unable to understand the consent/assent process and provide written informed consent;
2. are currently enrolled in another research study addressing HIV/STIs/PrEP;
3. participated in the IMARA-SA adaptation process. AGYW and FC must agree to participate as a dyad. AGYW refusal will supersede FC consent.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants will be eligible to participate if they are female.
Enrollment: 61 (Actual)
Dates: Start 2019-10-26 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geri R Donenberg, PhD, Principal Investigator — University of Illinois Chicago; Linda-Gail Bekker, MBChB, PhD, Principal Investigator — Desmond Tutu HIV Centre
Locations (1):
- Desmond Tutu HIV Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request, pending discussion with the study team about the planned use of the data.
Supporting Information: Study Protocol
Time Frame: Following all study publications

REFERENCES:
- [Derived] Merrill KG, Atujuna M, Emerson E, Blachman-Demner D, Bray BC, Bekker LG, Donenberg GR. Preliminary effectiveness and implementation outcomes of the IMARA-South Africa sexual health intervention on adolescent girls and young women: A pilot randomized trial. PLOS Glob Public Health. 2023 Feb 15;3(2):e0001092. doi: 10.1371/journal.pgph.0001092. eCollection 2023. PMID 36962830

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 dyads were enrolled. Two dyads were withdrawn due to ineligibility. A total of 118 participants (59 dyads) were allocated to either IMARA-SA or the Health Promotion Control Arm.
Period: Overall Study
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Started | 29 | 30
Number of Dyads Completing Intervention Day 1 | 26 | 28
Number of Dyads Completing Intervention Day 2 | 22 | 27
Number of AGYW Completing at Least One Primary Outcome Measure | 20 (Number of AGYW. Outcome data represents AGYW only.) | 19 (Number of AGYW. Outcome data represents AGYW only.)
Completed | 27 (Number of AGYW. Outcome data represents AGYW only.) | 24 (Number of AGYW. Outcome data represents AGYW only.)
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Population: Adolescent Girls and Young Women (AGYW, N=59) and Female Caregivers (FC, N=59) contributed data for Age, Sex, Region of Enrollment, Highest Education Achieved, and Supporting Self Financially variables. AGYW (N=59) contributed data for Type of Female Caregiver, Sexual Behavior, HIV Testing and Counseling, Sexually Transmitted Infections, Prescribed PrEP, and Adherence to PrEP variables.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Customized [Count of Participants; unit: Participants] — Population: AGYW contributed to AGYW Age data, N=59
  Participants
    AGYW Age: number analyzed (Participants) | 29 | 30 | 59
    AGYW Age: 15-17 years old | 17 | 17 | 34
    AGYW Age: 18-19 years old | 12 | 13 | 25
Age, Customized [Count of Participants; unit: Participants] — Population: FC contributed to FC Age data, N=59
  Participants
    FC Age: number analyzed (Participants) | 29 | 30 | 59
    FC Age: 24-29 years old | 11 | 6 | 17
    FC Age: 30-39 years old | 9 | 13 | 22
    FC Age: 40-49 years old | 7 | 7 | 14
    FC Age: 50 and older | 2 | 3 | 5
    FC Age: Missing Data | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 58 | 60 | 118
AGYW highest education achieved [Count of Participants; unit: Participants] — Population: AGYW contributed to AGYW highest education achieved data, N=59
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    Some or all of primary school | 11 | 11 | 22
    Some or all of secondary | 18 | 15 | 33
    Higher education | 0 | 4 | 4
FC highest education level acheived [Count of Participants; unit: Participants] — Population: FC contributed to FC highest education achieved data, N=59
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    No schooling | 3 | 2 | 5
    Some or all of primary school | 9 | 12 | 21
    Some or all of secondary | 13 | 12 | 25
    Higher education | 4 | 3 | 7
    Missing Data | 0 | 1 | 1
AGYW supported self financially in past year [Count of Participants; unit: Participants] — Population: AGYW contributed to AGYW supported self financially in past year data, N=59
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    (all) | 3 | 7 | 10
FC supported self financially in the past year [Count of Participants; unit: Participants] — Population: FC contributed to FC supported self financially in the past year data, N=59
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    (all) | 23 | 24 | 47
AGYW report of female caregiver participating [Count of Participants; unit: Participants] — Population: AGYW contributed to AGYW report of female caregiver participating data, N=59
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    Biological mother | 12 | 12 | 24
    Aunt | 6 | 10 | 16
    Sister | 7 | 4 | 11
    Cousin | 3 | 2 | 5
    Grandmother | 0 | 1 | 1
    Other | 1 | 1 | 2
Number of AGYW reporting ever had sex [Count of Participants; unit: Participants] — Sex is defined as vaginal or anal sex. Population: AGYW contributed to Number of AGYW reporting ever had sex data, N=59
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    (all) | 20 | 19 | 39
Number of AGYW who have had sex in past 6 months [Count of Participants; unit: Participants] — Population: Among AGYW who have ever had sex (n=39).
  Participants
    number analyzed (Participants) | 20 | 19 | 39
    (all) | 12 | 14 | 26
AGYW age at first sex [Mean (Standard Deviation); unit: years] — Population: Among AGYW who have ever had sex (n=39).
  years
    number analyzed (Participants) | 20 | 19 | 39
    (all) | 15.6 (1.10) | 15.7 (0.93) | 15.6 (1.01)
Number of AGYW reporting did not use a condom at last sex [Count of Participants; unit: Participants] — Population: Among AGYW who had sex in the past 6 months (n=26).
  Participants
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 4 | 7 | 11
Number of AGYW who report using condoms inconsistently in past 6 months [Count of Participants; unit: Participants] — Population: Among AGYW who had sex in the past 6 months (n=26).
  Participants
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 4 | 10 | 14
Number of AGYW who report using substances during sex in past 6 months [Count of Participants; unit: Participants] — Population: Among AGYW who had sex in the past 6 months (n=26).
  Participants
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 8 | 10 | 18
Number of AGYW who report 2 or more partners in the past 6 months [Count of Participants; unit: Participants] — Population: Among AGYW who had sex in the past 6 months (n=26).
  Participants
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 5 | 5 | 10
Number of AGYW Completing HIV Testing and Counseling (HTC) [Count of Participants; unit: Participants] — Population: Among AGYW who were not living with HIV at baseline (n=57).
  Participants
    number analyzed (Participants) | 29 | 28 | 57
    (all) | 28 | 28 | 56
Number of AGYW who tested positive for a Sexually Transmitted Infection (STI) [Count of Participants; unit: Participants] — Population: Among AGYW who completed STI testing (gonorrhea and/or chlamydia) at baseline (n=56).
  Participants
    number analyzed (Participants) | 28 | 28 | 56
    (all) | 12 | 9 | 21
Number of AGYW who were ever prescribed PrEP [Count of Participants; unit: Participants] — Population: AGYW contributed to Number of AGYW who were ever prescribed PrEP data, N=59
  Participants
    number analyzed (Participants) | 29 | 30 | 59
    (all) | 2 | 5 | 7
AGYW's Report of Adherence to PrEP [Mean (Standard Deviation); unit: score] — (0=low adherence to 100=high adherence)
  Scale is comprised of 3 items: number of days dose missed, how often did you take PrEP in the way you were supposed to, how good a job did you do at taking PrEP. Items were transformed to a 0-100 scale and averaged. Thirty was subtracted from number of days missed and multiplied by 3.33. Responses for remaining 2 items: never/very poor=0, rarely/poor=20, sometimes/fair=40, usually/good=60, almost always/very good=80, always/excellent=100. Population: Among AGYW who self-reported having ever been prescribed PrEP at baseline.
  score
    number analyzed (Participants) | 2 | 5 | 7
    (all) | 75.0 (14.9) | 69.1 (21.1) | 70.8 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of AGYW Who Tested Positive for a Sexually Transmitted Infection (STI)
Description: A positive test for at least one of two STIs: chlamydia and/or gonorrhea
Time Frame: 8-17 months post baseline
Population: Data represents AGYW. Denominator is those who completed STI testing at follow-up. Excludes one participant who completed STI testing at follow-up but did not receive STI treatment at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 18 | 16
Participants | 4 | 6
Statistical Analysis 1: Comparison: IMARA-SA Intervention Arm vs Health Promotion Control Arm; Test type: Superiority; p = 0.15, Regression, Logistic; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.04 to 1.59]

2. Primary Outcome: Number of AGYW Completing HIV Testing and Counseling (HTC)
Description: Completion of HIV Testing and Counseling (HTC)
Time Frame: 8-17 months post baseline
Population: Denominator is those who came to site for HTC at follow-up and were not living with HIV (39 came to site for follow-up, 2 were living with HIV and were removed).
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 20 | 17
Participants | 20 | 17

3. Primary Outcome: Number of AGYW Who Elected to Take Pre-Exposure Prophylaxis (PrEP)
Description: Uptake of Pre-Exposure Prophylaxis (PrEP) assessed as receipt of PrEP prescription from research team or other care provider after the baseline survey.
Time Frame: 8-17 months post baseline
Population: Denominator is those who completed follow-up surveys, were not living with HIV, and did not report having been prescribed PrEP at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 25 | 20
Participants | 17 | 9
Statistical Analysis 1: Comparison: IMARA-SA Intervention Arm vs Health Promotion Control Arm; Test type: Superiority; p = 0.10, Regression, Logistic; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.81 to 9.89]

4. Secondary Outcome: AGYW's Report of Adherence to PrEP
Description: Adherence to PrEP is measured using an adapted version of the Wilson scale (2017).
  Measure Description: (0=low adherence to 100=high adherence) Scale is comprised of 3 items: number of days dose missed, how often did you take PrEP in the way you were supposed to, how good a job did you do at taking PrEP.
  Items were transformed to a 0-100 scale and averaged. Thirty was subtracted from number of days missed and multiplied by 3.33. Responses for remaining 2 items: never/very poor=0, rarely/poor=20, sometimes/fair=40, usually/good=60, almost always/very good=80, always/excellent=100.
Time Frame: 6-10 months post baseline
Population: Denominator is those who reported being prescribed PrEP on the follow-up survey and not on the baseline survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 14 | 7
score on a scale | 60.7 (19.5) | 54.4 (30.8)
Statistical Analysis 1: Comparison: IMARA-SA Intervention Arm vs Health Promotion Control Arm; Test type: Superiority; p = 0.65, Regression, Linear; beta coefficient = 5.00, 95% CI 2-sided [-17.78 to 27.78]

5. Secondary Outcome: AGYW Condom Use at Last Sex
Description: Self-reported condom use at last vaginal or anal sex using the AIDS Risk Behavior Assessment (ARBA).
Time Frame: 6-10 months post baseline
Population: Denominator includes AGYW who reported sex in the past 6 months at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 18 | 9
Participants
  Yes | 10 | 4
  No | 8 | 5
Statistical Analysis 1: Comparison: IMARA-SA Intervention Arm vs Health Promotion Control Arm; Test type: Superiority; p = 0.70, Fisher Exact

6. Secondary Outcome: AGYW Consistency of Condom Use
Description: Self-reported consistency of condom use during vaginal and anal sex in the past 6-months using the AIDS Risk Behavior Assessment (ARBA).
Time Frame: 6-10 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 18 | 9
Participants
  Always | 10 | 4
  Less than always | 8 | 5
Statistical Analysis 1: Comparison: IMARA-SA Intervention Arm vs Health Promotion Control Arm; Test type: Superiority; p = .70, Fisher Exact

7. Secondary Outcome: AGYW Substance Use During Sex in the Past 6 Months
Description: Self-reported number of times had vaginal or anal sex while drinking or taking drugs in the past 6-months using the AIDS Risk Behavior Assessment (ARBA).
Time Frame: 6-10 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 18 | 9
Participants
  Never | 9 | 4
  1+ time | 9 | 5
Statistical Analysis 1: Comparison: IMARA-SA Intervention Arm vs Health Promotion Control Arm; Test type: Superiority; p = 1.00, Fisher Exact

8. Secondary Outcome: Number of Partners in the Past 6 Months
Description: Self-reported number of vaginal or anal sex partners in the past 6-months using the AIDS Risk Behavior Assessment (ARBA).
Time Frame: 6-10 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 18 | 9
Participants
  1 partner | 14 | 8
  2+ partners | 4 | 1
Statistical Analysis 1: Comparison: IMARA-SA Intervention Arm vs Health Promotion Control Arm; Test type: Superiority; p = 0.64, Fisher Exact

9. Other Pre Specified Outcome: Intervention Fidelity
Description: Number of IMARA intervention activities completed as planned.
Time Frame: Same day the IMARA intervention was conducted
Population: Proportion of IMARA intervention activities completed as planned. Fidelity was not measured for the health promotion control group. The number of units analyzed is the total number of activities in the IMARA intervention.
Measure: Number; unit: Number of IMARA intervention activities
Units Other Than Participants: Activities
Groups:
- IMARA Activities: Day 1 and Day 2 IMARA intervention activities across both AGYW and caregiver groups.
Arm/Group | IMARA Activities
Number analyzed (Participants) | 210
Number analyzed (Activities) | 210
Number of IMARA intervention activities | 199

10. Other Pre Specified Outcome: Intervention Reach
Description: The number of dyads who were eligible and consented/assented to participate in the study.
Time Frame: Enrollment
Population: Data represents number of dyads who were eligible and enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Participants: All study participants who were enrolled, completed baseline assessments, and were randomized.
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 59
Participants | 59

11. Other Pre Specified Outcome: Intervention Feasibility: Completed the First Intervention Day of IMARA
Description: The number of dyads in the IMARA-SA group who attend at least one IMARA-SA session
Time Frame: Baseline
Population: The number of dyads in the IMARA-SA group who attend at least one IMARA-SA session
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm
Number analyzed (Participants) | 29
Participants | 26

12. Other Pre Specified Outcome: Intervention Feasibility: Completed the Second Intervention Day of IMARA
Description: The number of dyads in the IMARA-SA group who attended the second IMARA-SA session
Time Frame: Baseline
Population: The number of dyads in the IMARA-SA group who attended the second IMARA-SA session
Measure: Count of Participants; unit: Participants
Arm/Group | IMARA-SA Intervention Arm
Number analyzed (Participants) | 29
Participants | 22

13. Other Pre Specified Outcome: Intervention Acceptability: How Knowledgeable Were Your Group Leaders About the Information Presented Today?
Description: Single item: How knowledgeable were your group leaders about the information presented today? Participants responded on a 1 (Not at all) to 5 (Extremely) scale. High scores indicate greater acceptability.
Time Frame: Immediately post-intervention Day 1 and Day 2
Population: 29 AGYW-FC dyads were randomized to IMARA-SA: 26 dyads completed Day 1 and 22 dyads completed Day 2. Data is missing for 6 AGYW who completed Day 1 and 1 FC who completed Day 2.
  30 AGYW-FC dyads were randomized to Health Promotion: 28 dyads completed Day 1 and 27 dyads completed Day 2. Data is missing for 2 AGYW and 3 FC who completed Day 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IMARA-SA Intervention Arm: The IMARA-SA intervention aligns with an ecological framework, emphasizing the intersection of individual, social, and structural determinants of women's sexual health and behavior. Separate FC and AGYW groups run simultaneously and cover parallel content, while joint activities enhance FC credibility as a resource for HIV/STI prevention and facilitate practice of communication skills. Interventionists use interactive and experiential activities. IMARA-SA's goals and motto emphasize strong FC-AGYW relationships, sisterhood, community empowerment, and motivation for HIV prevention, and build group cohesion. FC and AGYW sign a pact to confirm commitment to the program. At the end of Workshop Day 1, participants receive homework to complete during the week. Woven throughout IMARA-SA is the impact of mental health issues, alcohol and drug use, and violence on HIV-risk.
- Health Promotion Control Arm: The health promotion control intervention is a family-based intervention previously delivered tofamilies in SA and translated into isiXhosa. The intervention promotes healthy living by encouraging good nutrition,exercise, and violence reduction. It is delivered in the same format as IMARA and is identical in length and intensity.
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 58 | 60
units on a scale
  AGYW Day 1: number analyzed (Participants) | 20 | 28
  AGYW Day 1 | 4.90 (.31) | 4.86 (.45)
  FC Day 1: number analyzed (Participants) | 26 | 28
  FC Day 1 | 4.88 (.33) | 4.75 (.59)
  AGYW Day 2: number analyzed (Participants) | 22 | 25
  AGYW Day 2 | 4.73 (.55) | 4.80 (.41)
  FC Day 2: number analyzed (Participants) | 21 | 24
  FC Day 2 | 4.86 (.36) | 4.88 (.34)

14. Other Pre Specified Outcome: Intervention Acceptability: How Satisfied Were You With Today's Workshop?
Description: Single item: How satisfied were you with today's workshop? Participants responded on a 1 (Not at all) to 5 (Extremely) scale. High scores indicate greater acceptability.
Time Frame: Immediately post-intervention Day 1 and Day 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Health Promotion Control Arm: The health promotion control intervention is a family-based intervention previously delivered to families in SA and translated into isiXhosa. The intervention promotes healthy living by encouraging good nutrition, exercise, and violence reduction. It is delivered in the same format as IMARA and is identical in length and intensity.
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 58 | 60
units on a scale
  AGYW Day 1: number analyzed (Participants) | 20 | 28
  AGYW Day 1 | 4.95 (.22) | 4.54 (.69)
  FC Day 1: number analyzed (Participants) | 26 | 28
  FC Day 1 | 4.85 (.37) | 4.79 (.50)
  AGYW Day 2: number analyzed (Participants) | 22 | 25
  AGYW Day 2 | 4.86 (.35) | 4.80 (.58)
  FC Day 2: number analyzed (Participants) | 21 | 24
  FC Day 2 | 4.76 (.44) | 5.00 (.00)

15. Other Pre Specified Outcome: Intervention Acceptability: How Comfortable Were You With the Group Leaders Who Worked With You Today?
Description: Single item: How comfortable were you with the group leaders who worked with you today? Participants responded on a 1 (Not at all) to 5 (Extremely) scale. High scores indicate greater acceptability.
Time Frame: Immediately post-intervention Day 1 and Day 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 58 | 60
units on a scale
  AGYW Day 1: number analyzed (Participants) | 20 | 28
  AGYW Day 1 | 4.65 (.49) | 4.89 (.32)
  FC Day 1: number analyzed (Participants) | 26 | 28
  FC Day 1 | 4.73 (.53) | 4.79 (.50)
  AGYW Day 2: number analyzed (Participants) | 22 | 25
  AGYW Day 2 | 4.68 (.57) | 4.80 (.41)
  FC Day 2: number analyzed (Participants) | 21 | 24
  FC Day 2 | 4.90 (.30) | 4.96 (.20)

16. Other Pre Specified Outcome: Intervention Acceptability: How Much Did You Feel the Group Leaders Valued What You Said?
Description: Single item: How much did you feel the group leaders valued what you said? Participants responded on a 1 (Not at all) to 5 (Extremely) scale. High scores indicate greater acceptability.
Time Frame: Immediately post-intervention Day 1 and Day 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 58 | 60
units on a scale
  AGYW Day 1: number analyzed (Participants) | 20 | 28
  AGYW Day 1 | 4.75 (.55) | 4.79 (.42)
  FC Day 1: number analyzed (Participants) | 26 | 28
  FC Day 1 | 4.88 (.33) | 4.79 (.57)
  AGYW Day 2: number analyzed (Participants) | 22 | 25
  AGYW Day 2 | 4.68 (.57) | 4.76 (.44)
  FC Day 2: number analyzed (Participants) | 21 | 24
  FC Day 2 | 4.95 (.22) | 4.88 (.34)

17. Other Pre Specified Outcome: Intervention Acceptability: How Honest Did You Feel You Could be During Today's Workshop?
Description: Single item: How honest did you feel you could be during today's workshop? Participants responded on a 1 (Not at all) to 5 (Extremely) scale. High scores indicate greater acceptability.
Time Frame: Immediately post-intervention Day 1 and Day 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 58 | 60
units on a scale
  AGYW Day 1: number analyzed (Participants) | 20 | 28
  AGYW Day 1 | 4.70 (.57) | 4.64 (.56)
  FC Day 1: number analyzed (Participants) | 26 | 28
  FC Day 1 | 4.69 (.62) | 4.82 (.39)
  AGYW Day 2: number analyzed (Participants) | 22 | 25
  AGYW Day 2 | 4.73 (.55) | 4.80 (.50)
  FC Day 2: number analyzed (Participants) | 21 | 24
  FC Day 2 | 4.86 (.36) | 5.00 (.00)

18. Other Pre Specified Outcome: Intervention Acceptability: How Much Did You Feel You Were Involved or Engaged in the Activities?
Description: Single item: How much did you feel you were involved or engaged in the activities? Participants responded on a 1 (Not at all) to 5 (Extremely) scale. High scores indicate greater acceptability.
Time Frame: Immediately post-intervention Day 1 and Day 2
Population: 29 AGYW-FC dyads were randomized to IMARA-SA: 26 dyads completed Day 1 and 22 dyads completed Day 2. Data is missing for 6 AGYW who completed Day 1, 1 AGYW who completed Day 2, and 1 FC who completed Day 2.
  30 AGYW-FC dyads were randomized to Health Promotion: 28 dyads completed Day 1 and 27 dyads completed Day 2. Data is missing for 2 AGYW and 3 FC who completed Day 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
Number analyzed (Participants) | 58 | 60
units on a scale
  AGYW Day 1: number analyzed (Participants) | 20 | 28
  AGYW Day 1 | 4.75 (.44) | 4.71 (.60)
  FC Day 1: number analyzed (Participants) | 26 | 28
  FC Day 1 | 4.58 (.64) | 4.68 (.61)
  AGYW Day 2: number analyzed (Participants) | 21 | 25
  AGYW Day 2 | 4.67 (.58) | 4.72 (.54)
  FC Day 2: number analyzed (Participants) | 21 | 24
  FC Day 2 | 4.95 (.22) | 4.75 (.61)

ADVERSE EVENTS:
Time Frame: Data were collected from enrollment to follow-up visit (8 to 17 months post baseline).
Arm/Group | IMARA-SA Intervention Arm | Health Promotion Control Arm
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT05504954/Prot_SAP_000.pdf
  • Informed Consent Form: ICF for Girls between the ages of 18-19 (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05504954/ICF_001.pdf
  • Informed Consent Form: Parent ICF for Minors (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05504954/ICF_002.pdf
  • Informed Consent Form: ICF for Caregiver's own participation (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05504954/ICF_003.pdf
  • Informed Consent Form: Assent for Minors (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05504954/ICF_004.pdf